CLINICAL TRIAL: NCT04568928
Title: Implementation of Locomotor Training Program Using a Powered Exoskeleton Combined With Functional Electrical Stimulation in Clinical Practice for Persons With an Incomplete Spinal Cord Injury - WHY and HOW to do it?
Brief Title: Powered Exoskeleton Combined With Functional Electrical Stimulation in Clinical Practice
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Laval University (Other)
Collaborators: Praxis Spinal Cord Institute (Other)
Responsible Party: Principal Investigator, François Routhier, Full Professor/ Researcher, Laval University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-2002
Record Dates: First submitted 2020-09-11; First posted 2020-09-29 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Incomplete Spinal Cord Injury
Keywords: Exoskeleton, locomotor training, FES, SCI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OLTP/PE+FES (Experimental): 3-5 familiarization sessions + 12 training sessions (3 blocks of 4 training sessions; 60-90 min each session, 2-3 sessions per week) of an overground locomotor training program using a powered exoskeleton combined with functional electrical stimulation (OLTP/PE+FES).
  The training sessions are divided into 3 blocks. Each block will take place over a period of approximately 2 weeks (2-3 sessions/week) and will consist of 3 training sessions with exoskeleton combined with FES and a fourth session with exoskeleton alone, without FES.
  For each participant, FES intensity will be set for each muscle in order to elicit a palpable muscle contraction. FES timing and duration is already built into the device. For each participant, specific level of assistance for each hip and knee, and gait parameters will be set and adjusted during a familiarization period with the PE. Level of PE assistance will then be adjusted weekly to ensure training progression.
  Interventions: Device: OLTP/PE + FES

INTERVENTIONS:
Device: OLTP/PE + FES — 12 sessions OLTP/PE + FES

SUMMARY:
After partial spinal cord injury, gait deficits may be present and often remain even after intensive rehabilitation. New robotic technologies have recently emerged to help augment the extent of rehabilitation. However, these are complex tools to integrate into clinical practice and little is known about the potential factors that may influence the uptake of a locomotor program using this technology by clinicians. The goal of this project is to bring together researchers, administrators, clinicians and patients to define and implement an overground robotized gait training program in clinic. We will also investigate the added value of leg and trunk muscle stimulation combined with robotic walking training, to see if it could enhance recovery.

DETAILED DESCRIPTION:
Powered exoskeleton technology represents a promising rehabilitation intervention for persons with incomplete spinal cord injury (iSCI). The overall aim of the present study is to investigate the implementability of an overground locomotor training program using a powered exoskeleton in persons with a subacute iSCI at the Institut de réadaptation en déficience physique de Québec, with and without functional electrical stimulation (FES). Over the 2-year period of the project, a logic model will be co-developed with stakeholders to support clinicians and administrators in the management of the locomotor training program. Using qualitative and quantitative research methods, we will evaluate the feasibility and perceived barriers/facilitators to the implementation in clinical practice of the training program. Finally, a pre-post design with individuals receiving the intervention either combined with FES or not, will allow quantifying of the benefits of combining FES in addition to robotic gait training on functional walking capacity in persons with a subacute iSCI.

ELIGIBILITY:
Inclusion Criteria:

General

* Measure between 5'1" and 6'3" (1.5 and 1.9m)
* Weigh less than 200 pounds (90kg)
* Present a diagnosis of incomplete spinal cord injury
* Have the ability to maintain a standing position and/or have therapeutic walking ability at Stage 1B or more of the Rick Hansen Institute SCI Standing and Walking Assessment Toolkit
* Present sufficient upper extremity strength and function to use a walker with wheels
* Femur length between 37 and 49cm
* Width of hips when seated <42 cm
* Obtain approval from a physician to participate in the project
* Standing tolerance >15 minutes

For FES:

* Respond favourably to functional electrical stimulation (FES) of the main lower extremity muscle groups: (gluteus, quadriceps, hamstrings, dorsiflexors, etc.) as determined by a physiotherapist.
* Have no contraindications to FES according to the guidelines of the Canadian physiotherapy association (CPA).

Exclusion Criteria:

General:

* Poor fit of the exoskeleton as determined by the research team
* Present contraindications to the use of the Indego® exoskeleton as described by the company
* Present lower extremity skin lesions or sores
* Any medical condition or co-morbidity that may impair collaboration and participation or making it unsafe to wear the exoskeleton, for example (non-exhaustive list) :
* Disabling pain.
* Significant sensory disturbances in the lower limbs that limit safe walking.
* Cognitive disorders that impair the ability to collaborate.
* Osteoporosis.
* Unconsolidated fractures of the lower limbs.
* Uncontrolled reflex dysautonomia.
* Severe peripheral vascular disease.
* Severe heart failure.
* Severe, active infection

FES Exclusion Criteria

* Pregnancy;
* Presence of a malignant tumor
* Deep vein thrombosis
* Hemorrhagic condition
* Infection or osteomyelitis
* Presence of weakened/damaged skin
* Circulatory disorders
* Epilepsy
* Electronic implant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-12-10 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Change in Modified Six Minute Walk Test (6MWT) | 2 assessment timepoints: at baseline, at the end of the intervention (1 to 2 weeks later)
  A walking endurance test that measures the longest distance covered continuously during a maximum of six minutes.
Change in 10 meter Walk Test (10mWT) | 2 assessment timepoints: at baseline, at the end of the intervention (1 to 2 weeks later)
  Measures preferred and maximal walking speeds over 10 meters
Change in Modified Timed Up and Go test (TUG) | 2 assessment timepoints: at baseline, at the end of the intervention (1 to 2 weeks later)
  A functional test that assesses sit-to-stand transfers, balance and mobility
Change in Walking Index for Spinal Cord Injury (WISCI-II) | 2 assessment timepoints: at baseline, at the end of the intervention (1 to 2 weeks later)
  functional walking capacity scale that describes the amount of physical assistance, braces or devices required to walk 10 meters

SECONDARY OUTCOMES:
Change in Brief pain inventory questionnaire | 2 assessment timepoints: at baseline, at the end of the intervention (1 to 2 weeks later)
  Intensity of pain
Change in Spinal Cord Injury Secondary Conditions scale (SCI-SCS) | 2 assessment timepoints: at baseline, at the end of the intervention (1 to 2 weeks later)
  This scale specifically targets secondary conditions associated with SCI that directly and indirectly impact health and physical functioning. The rating scale uses a 4-point ordinal scale ranging from 0 (not experienced/insignificant problem never limiting activity) to 3 (significant/chronic problem). Total scores range from 0 to 48. Higher scores indicate greater overall problems with secondary conditions
Change in the Modified Ashworth Scale (MAS) | 2 assessment timepoints: at baseline, at the end of the intervention (1 to 2 weeks later)
  A measure of lower limb spasticity. Scores range from 0 to 4. Higher scores indicate greater spasticity.
  scale.
Change in electromyographic (EMG) activity of the tibialis anterior, triceps surae, quadriceps, hamstrings muscles during walking.will be recorded using a Delsys Trigno system. | 2 assessment timepoints: at baseline, at the end of the intervention (1 to 2 weeks later)
  Muscle activation patterns (i.e., amplitude, timing) and muscle fatigue (reduction in the median frequency of the EMG power spectrum) will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: François Routhier, PhD, Principal Investigator — Laval University
Locations (1):
- Laval University, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided